CLINICAL TRIAL: NCT01123187
Title: Phase 2 Study of Islet Cell Transplantation in Patients With Type I Diabetes With Previous Kidney Transplantation With Steroid Free Immunosuppression
Brief Title: Islet Cell Transplantation in Patients With Type I Diabetes With Previous Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 95/120; 98001 (Other: Sponsor); DGS 980032 (Other: AFSSAPS)
Record Dates: First submitted 2010-05-11; First posted 2010-05-14 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes; Organ Transplantation; Immunosuppression
Keywords: diabetes type 1; kidney transplantation; islet; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Intervention Model Description: Islet transplantation
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- islet transplantation (Experimental): Islet transplantation
  Interventions: Procedure: islet transplantation

INTERVENTIONS:
Procedure: islet transplantation — Islet transplantation consisted of up to three sequential fresh islet infusions within three months. Access to the portal vein was gained under general anesthesia by percutaneous catheterisation of a peripheral portal branch under ultrasound guidance or by surgical catheterisation of a small mesenteric vein.
  Other Names: surgical catheterisation; percutaneous catheterisation

SUMMARY:
This single center phase 2 clinical trial, is designed for confirming the efficacy and safety of sequential islet allotransplantation with steroid free immunosuppression in patients with previous kidney transplantation.

DETAILED DESCRIPTION:
The beneficial effects of glycemic control on both survival and function of transplanted kidneys in patients with type 1 diabetes mellitus have been recognized.

The purpose of this study is to reverse hyperglycemia and insulin dependency, by islet cell transplantation, in patients with type 1 diabetes mellitus who have a stable kidney allograft.

The study primary efficacy endpoint is graft survival defined as insulin independence and HbA1c < 8% at 1 year post first transplant. Secondary outcomes are graft function and metabolic control

The immunosuppression protocol for the kidney graft was converted to sirolimus+tacrolimus regimen 6 months before islet transplantation to exclude negative effects on kidney graft function.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus. Documentation of negative basal and stimulated C-peptide and diagnosis of diabetes for at least 5 years.
* Recipient of renal transplant with good function (creatinine clearance >/=60 ml/min)
* Stable immunosuppression consisting of any combination of sirolimus, tacrolimus for at least 6 months, without major complications
* Ability to give informed consent.
* Age greater than or equal to 18 years or less than or equal to 65 years
* No evidence of liver disease (liver enzymes < twice the upper limit of normal)

Exclusion Criteria:

* Age below 18 years and above 65 years
* Significant cardiovascular disease, including non-correctable coronary artery disease and/or recent myocardial infarction(within last 12 months); extensive peripheral vascular disease not correctable by surgery, unstable angina
* Untreated proliferative retinopathy.
* Recent Cerebrovascular accident (within last 12 months)
* Recent unresolved acute infection, or chronic infection, including tuberculosis, HIV, HBV, HCV, CMV or positive skin test for TB
* Any history of malignancy, except squamous or basal skin cancer or in situ cancer of the cervix.
* History of non-compliance, or inability to demonstrate capacity to comply with strict blood glycemic control and insulin pump therapy.
* Psychiatric illness that is untreated, or likely to interfere significantly with transplantation despite treatment.
* Pregnant women, women intending future pregnancy, women of reproductive potential who are unable or unwilling to follow effective contraceptive measures for the duration of immunosuppressive therapy
* Fasting C-peptide > 0.2 ng/ml
* Creatinine > 25mg/l
* Alkaline phosphatase, total bilirubin, Alanine Aminotransferase (ALT)or Aspartate Aminotransferase (AST) > twice the upper limit of normal
* Significant liver disease (elevation of liver enzymes > twice the upper limit of normal for each of ALT and AST, liver masses including portal vein thrombosis, evidence of portal hypertension, or significant, untreated gallbladder disease (i.e., gallstones).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2003-03; Primary Completion 2014-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Composite criteria: insulin independence and Glycosylated Hemoglobin (HbA1c) under 8% at one year after the transplantation | One year
  Percent of insulin-independent patients with a Glycosylated Hemoglobin (HbA1c) under 8% at one year after injection of approximately 10,000 islets equivalents / kg (IE/kg).

SECONDARY OUTCOMES:
The number of adverse events | 1 year
  The number of adverse events related to the procedure and to the immunosuppression
Number of severe episodes of hypoglycemia | 1 year
  Number of severe episodes of hypoglycemia (requiring the use of third)
Evaluation of Diabetes complications | 1 year
  Evaluation of Diabetes complications: retinopathy, neuropathy, nephropathy
Lipid metabolism | 1 year
  Lipid metabolism assessed by measurement of total cholesterol and HDL cholesterol, triglycerides, ApoA1, apoB, apoE, free fatty acids and lipid.
Evaluation of kidney function | 1 year
  Evaluation of kidney function (creatinine, creatinine clearance,proteinurie)

CONTACTS AND LOCATIONS:
Overall Officials: François PATTOU, MD, PhD, Principal Investigator — University Hospital, Lille; Marie-Christine VANTYGHEM, MD, Principal Investigator — University Hospital, Lille; Christian NOEL, MD, Principal Investigator — University Hospital, Lille; Julie KERR-CONTE, MD, Principal Investigator — Université de Lille 2
Locations (1):
- University Hospital of Lille, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vantyghem MC, Kerr-Conte J, Arnalsteen L, Sergent G, Defrance F, Gmyr V, Declerck N, Raverdy V, Vandewalle B, Pigny P, Noel C, Pattou F. Primary graft function, metabolic control, and graft survival after islet transplantation. Diabetes Care. 2009 Aug;32(8):1473-8. doi: 10.2337/dc08-1685. PMID 19638525
- [Derived] Vantyghem MC, Chetboun M, Gmyr V, Jannin A, Espiard S, Le Mapihan K, Raverdy V, Delalleau N, Machuron F, Hubert T, Frimat M, Van Belle E, Hazzan M, Pigny P, Noel C, Caiazzo R, Kerr-Conte J, Pattou F; Members of the Spanish Back Pain Research Network Task Force for the Improvement of Inter-Disciplinary Management of Spinal Metastasis. Ten-Year Outcome of Islet Alone or Islet After Kidney Transplantation in Type 1 Diabetes: A Prospective Parallel-Arm Cohort Study. Diabetes Care. 2019 Nov;42(11):2042-2049. doi: 10.2337/dc19-0401. PMID 31615852
- [Derived] Benomar K, Chetboun M, Espiard S, Jannin A, Le Mapihan K, Gmyr V, Caiazzo R, Torres F, Raverdy V, Bonner C, D'Herbomez M, Pigny P, Noel C, Kerr-Conte J, Pattou F, Vantyghem MC. Purity of islet preparations and 5-year metabolic outcome of allogenic islet transplantation. Am J Transplant. 2018 Apr;18(4):945-951. doi: 10.1111/ajt.14514. Epub 2017 Nov 11. PMID 28941330
- [Derived] Caiazzo R, Vantyghem MC, Raverdi V, Bonner C, Gmyr V, Defrance F, Leroy C, Sergent G, Hubert T, Ernst O, Noel C, Kerr-Conte J, Pattou F. Impact of Procedure-Related Complications on Long-term Islet Transplantation Outcome. Transplantation. 2015 May;99(5):979-84. doi: 10.1097/TP.0000000000000458. PMID 25393157
- [Derived] Vantyghem MC, Raverdy V, Balavoine AS, Defrance F, Caiazzo R, Arnalsteen L, Gmyr V, Hazzan M, Noel C, Kerr-Conte J, Pattou F. Continuous glucose monitoring after islet transplantation in type 1 diabetes: an excellent graft function (beta-score greater than 7) Is required to abrogate hyperglycemia, whereas a minimal function is necessary to suppress severe hypoglycemia (beta-score greater than 3). J Clin Endocrinol Metab. 2012 Nov;97(11):E2078-83. doi: 10.1210/jc.2012-2115. Epub 2012 Sep 20. PMID 22996144